CLINICAL TRIAL: NCT06892015
Title: OBSERVATIONAL STUDY ON VIRAL SHEDDING AND IMMUNOLOGICAL RESPONSE OF OROPOUCHE VIRUS
Acronym: OROVIMM
Status: Recruiting | Type: Observational
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-ZN
Record Dates: First submitted 2025-03-10; First posted 2025-03-24 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Oropouche Infection
MeSH Terms: conditions — Bunyaviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — The following clinical specimens will be collected:
  1. Urine (10mL)
  2. Whole Blood (EDTA tube 2x7mL)
  3. Serum (2x7mL)
  4. CSF (1mL) - only if the physician requires this sampling as per normal clinical practice, based on the patient's clinical presentation
  5. Amniotic fluid (5mL) - only if the physician requires this sampling as per normal clinical practice, based on the patient's clinical presentation
  6. Seminal fluid (1mL) - this sample is not mandatory, we will collect them only from subjects agreeing to donate.
  7. Vaginal swab in UTM medium - this sample is not mandatory, we will collect them only from subjects agreeing to donate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OROV patients: The study population will consist of adult patients (age 18 years or over) with RT-PCR-confirmed OROV, who attended or will attend health services at DITM. During first clinical encounter, study participants will be interviewed and physically examined as part of routine clinical practice, in this occasion patients will be also approached to obtain informed consent by their attending physician; all the patients will also be asked the consent for the donation of residual samples from routine diagnostic tests to Tropica BioBank.
  RT-PCR and culture testing will be repeated at each clinical visit and will stop when one negative RT-PCR results from all matrices have been obtained. Immunologic testing will continue for the duration of the study.
  Subject participation duration will be about 3 months in total.

SUMMARY:
This is a single-center observational study, whose primary objective is to describe the immune response to Oropouche Virus (OROV) during the study period and the duration of viral RNA shedding, only for sequential samples, by RT-PCR in different matrices.

DETAILED DESCRIPTION:
This is a study with retrospective and prospective enrollment.

ELIGIBILITY:
Inclusion Criteria:

* patients resulted positive to the RT-PCR for OROV;
* informed consent to the participation to the study and to personal data's treatment and/or donation of residual samples to Tropika Biobank;
* patients ≥ 18 years old.

Exclusion Criteria

• lack of signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (age 18 years or over) with RT-PCR-confirmed OROV, who attended or will attend health services at the Center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Anti-OROV serum antibody response | Baseline, 7 days post symptoms onset (DPSO), 14 days DPSO, 21 days DPSO, 28days DPSO, 60days DPSO, 90days DPSO
  Results of the anti-OROV serum antibody response along the study period:
  * IgM (titer, reciprocal of dilution);
  * IgG (titer, reciprocal of dilution).
OROV viral RNA shedding in different matrices | Baseline, 7 days post symptoms onset (DPSO), 14 days DPSO, 21 days DPSO, 28days DPSO, 60days DPSO, 90days DPSO
  Results of OROV viral RNA presence in different matrice along the study period:
  RT-PCR Ct and RNA copies/mL in different matrices: urine, whole blood, serum, vaginal swab or seminal fluid, CSF and amniotic fluid if available.

SECONDARY OUTCOMES:
Quality of anti-OROV humoral response | Baseline, 7 days post symptoms onset (DPSO), 14 days DPSO, 21 days DPSO, 28days DPSO, 60days DPSO, 90days DPSO.
  Results of the anti-OROV neutralizing antibody response along the study period:
  neutralizing antibodies titer (titer, reciprocal of dilution).
Quality of anti-OROV cell mediated immunity evolution | Baseline, 7 days post symptoms onset (DPSO), 14 days DPSO, 21 days DPSO, 28days DPSO, 60days DPSO, 90days DPSO
  Results of the quality of anti-OROV cell mediatedimmune response along the study period: specific cell-mediated response (specific IFN producing cells/100,000).
Quality of anti-OROV cytokine production | Baseline, 7 days post symptoms onset (DPSO), 14 days DPSO, 21 days DPSO, 28days DPSO, 60days DPSO, 90days DPSO.
  Results of the quality of anti-OROV cytokine production profile along the study period: cytokine analysis (pg/ml)
Timing evolution of humoral OROV specific response | Baseline, 7 days post symptoms onset (DPSO), 14 days DPSO, 21 days DPSO, 28days DPSO, 60days DPSO, 90days DPSO
  IgM and IgG kinetics (days from symptoms onset or first diagnosis).
Time duration limits of RT-PCR-positivity persistence in different matrices | Baseline, 7 days post symptoms onset (DPSO), 14 days DPSO, 21 days DPSO, 28days DPSO, 60days DPSO, 90days DPSO
  RT-PCR positivity persistence (days from symptoms onset or first diagnosis)
Semi-quantitative OROV RNA viral loads evaluation | Baseline, 7 days post symptoms onset (DPSO), 14 days DPSO, 21 days DPSO, 28days DPSO, 60days DPSO, 90days DPSO
  Results of OROV RT-PCR testing results by cycle threshold (Ct) values along the study period: RT-PCR (Ct)
Quantitative OROV RNA viral load evaluation | Baseline, 7 days post symptoms onset (DPSO), 14 days DPSO, 21 days DPSO, 28days DPSO, 60days DPSO, 90days DPSO
  Results of OROV RNA copies along the study period: ddPCR (copies/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria, Negrar, VR, Italy